CLINICAL TRIAL: NCT00837395
Title: Inflammatory Mediators and microRNA Analysis in Premenstrual Asthma
Status: Terminated | Type: Observational
Why Stopped: Co-investigator left the university and another co-investigator died several years ago, making it impossible to complete the study as planned.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jennifer McCallister MD, Associate Professor Clinical Internal Medicine, Ohio State University
Other Study IDs: 2008H0292
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Asthma
Keywords: premenstrual increase in asthma symptoms
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- premenstual asthma: women with asthma have an increase in asthma symptoms during the premenstrual or menstrual period

SUMMARY:
A small number of women with asthma have an increase in asthma symptoms during the premenstrual or menstrual period. This study is being done to investigate the possible causes of this premenstrual increase in asthma symptoms and to help asthma care providers identify those patients who may suffer from this condition.

DETAILED DESCRIPTION:
It is well established that women suffer more asthma symptoms and worse health-related quality of life than men with the same level of asthma severity. The etiology for these sex-related differences in unknown, but a subset of women has premenstrual asthma (PMA) with worsening of their asthma symptoms either prior to or during menstruation. Previous small trials have suggested that an increase in the host inflammatory response may correlate with PMA symptoms. We have evidence that small inhibitory ribonucleic acids, microRNAs, circulating in the peripheral blood of human patients may be expressed in different patterns in certain disease states when compared to healthy individuals.

We plan to compare the patterns of microRNA expression in a well characterized group of women with PMA to those without PMA to determine if alterations in these microRNA patterns play a role in increased asthma symptoms in the premenstrual period. In addition, we plan to compare the levels of inflammatory markers in these populations to better define the specific subset of women that may be at risk for premenstrual asthma. By better characterizing these women, we hope to identify clinically relevant predictors that may guide therapy for women who suffer from PMA.

Procedures to be used in this study include questionnaire administration, pulmonary function assessment, exhaled nitric oxide evaluation, urine sampling for pregnancy, and blood draws for microRNA and serum leukotriene evaluation. These techniques are utilized widely in clinical asthma research, and are associated with minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma

Exclusion Criteria:

* Are pregnant
* Take hormonal medication
* Have an illness with fever (> 38.0 ˚ C or 100.4 ˚ F) within 24 hours of Visit 1 or between Visits 1 and 2
* Are participating in another interventional research trial
* Have other major chronic illnesses that would interfere with participation
* Are taking the following medications: leukotriene receptor antagonists, oral steroids, anticoagulants, or insulin
* Are unable to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
To determine the patterns of serum microRNA in asthmatic women with premenstrual asthma and asthmatic women without premenstrual asthma at baseline and during the premenstrual period | during the study
  microRNA patterns in women with premenstrual asthma

SECONDARY OUTCOMES:
To determine the level of exhaled nitric oxide and serum leukotrienes B4 (LTB4) and C4 (LTC4) in asthmatic women with premenstrual asthma and asthmatic women without premenstrual asthma at baseline and during the premenstrual period | during the study
  Inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McCallister, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States